CLINICAL TRIAL: NCT05566379
Title: Effects of a Mindfulness Intervention on Physical and Psychological Well-Being and Quality of Life in Patients With Post Acute Sequelae of SARS-CoV-2 Infection (PASC) Dysautonomia
Brief Title: Mindfulness in Post Acute Sequelae of SARS-CoV-2 Infection (PASC) Dysautonomia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Jeffrey J. Hsu, Principal Investigator, University of California, Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 22-001020
Record Dates: First submitted 2022-10-02; First posted 2022-10-04 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-06

CONDITIONS: Long COVID; Dysautonomia
Keywords: Mindfulness , Long COVID, Dysautonomia
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome; Autonomic Nervous System Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mindfulness Intervention (Experimental): All participants will attend a virtual 6-week course entitled Mindful Awareness Practices (MAPs) created, hosted and led by expert facilitators from the Mindful Awareness Research Center at UCLA. Participants will learn Mindful concepts and a variety of Mindfulness practices. This intervention will consist of a mix of lecture, practice, group feedback, and discussion regarding mindfulness. Mindfulness is the mental state achieved by focusing one's awareness on the present while acknowledging and accepting any feelings, thoughts, or bodily sensations. MAPs classes meets weekly for two hours per week for six weeks. Participants are encouraged to complete some daily meditation practice starting at five minutes a day and working up to 20 minutes daily by the end of the course.
  Interventions: Other: Mindfulness - Mindful Awareness Practices ( MAPs)

INTERVENTIONS:
Other: Mindfulness - Mindful Awareness Practices ( MAPs) — All participants will attend a virtual 6-week course entitled Mindful Awareness Practices (MAPs) created, hosted and led by expert facilitators from the Mindful Awareness Research Center at UCLA. Participants will learn Mindful concepts and a variety of Mindfulness practices. This intervention will consist of a mix of lecture, practice, group feedback, and discussion regarding mindfulness. Mindfulness is the mental state achieved by focusing one's awareness on the present while acknowledging and accepting any feelings, thoughts, or bodily sensations. MAPs classes meets weekly for two hours per week for six weeks. Participants are encouraged to complete some daily meditation practice starting at five minutes a day and working up to 20 minutes daily by the end of the course.

SUMMARY:
The current pilot study will recruit participants experiencing new, returning, or ongoing symptoms related to COVID-19 illness for at least four weeks after being first infected with SARS-CoV-2. All participants will attend a virtual 6-week course entitled Mindful Awareness Practices (MAPs) created, hosted and led by expert facilitators from the Mindful Awareness Research Center (MARC) at University of California Los Angeles (UCLA). This intervention will consist of a mix of lecture, practice, group feedback, and discussion regarding mindfulness. Mindfulness is the mental state achieved by focusing one's awareness on the present while acknowledging and accepting any feelings, thoughts, or bodily sensations. The research team will collect self-reported measures of mental health symptoms, physical health symptoms, and demographic information before and after participants attend MAPs. Objective health measures will also be collected by the research team including an active stand test, a 6-minute walk, and a blood sample.

DETAILED DESCRIPTION:
The purpose of the current pilot project is to assess the feasibility and effects of a 6-week group mindfulness intervention in patients with Post Acute Sequelae of SARS-CoV-2 Infection (PASC)-related dysautonomia.

This single-arm study uses a one group pretest/posttest design. A convenience sample of patients will be recruited from the Ahmanson-University of California Los Angeles (UCLA) COVID-19 Cardiology Specialty Clinic and UCLA Long COVID Program.

Outcomes Measures:

Once consented, eligible participants will complete a baseline demographics survey, preintervention assessments including the composite autonomic symptom scoring (COMPASS-31), outcome measures questionnaires for perceived stress, anxiety, depression, fatigue, resilience, sleep, event specific distress, well-being and quality of life. A peripheral blood collection device for evaluation of inflammatory gene expression will be performed along with an active stand test and 6- minute walk prior to the mindfulness intervention. The same measures will be collected following completion of the intervention. Additionally, a logbook of patient self-reported practice frequency will be reviewed, and a focused 3 question audio recorded interview will be conducted at the post intervention visit. At 4-week follow-up post intervention, the final set of assessment questionnaires, and a 3-question mindfulness experience survey will be collected.

Intervention:

Participants will complete a virtual group based 6-week mindfulness meditation-based intervention, Mindful Awareness Practices (MAPs), developed by Diana Winston and colleagues at the Mindful Awareness Research Center (MARC) at UCLA. In response to COVID-19 precautions participants will meet virtually for six weekly, 2-hour group sessions. The group size is estimated at 15 participants.

MAPs is a standardized intervention that has been used in several previous studies. MAPS includes presentation of theoretical framework and materials on mindfulness, relaxation, and the mind-body connection, and experiential practice of meditation. Lecture, discussion, and group process focus on solving problems concerning barriers to effective practice, working with difficult thoughts and emotions, managing pain, and cultivation of loving kindness. Written materials are provided with a summary of information covered each week. Additionally, participants are instructed to practice mindfulness exercises at home on a daily basis (5-20 minutes/day) and advised in the informal use of mindfulness in daily life. Participants will be asked to keep a self-reported log of their daily practice. Classes will be led by experienced mindfulness instructors who received specialized training at the UCLA MARC Center.

Overview:

Baseline Visit (in person): collect within 1-2 week(s) prior to the intervention.

Consent Baseline demographics survey COMPASS-31: the composite autonomic symptom score Questionnaires: perceived stress (PSS), anxiety (GAD-7), depression (PHQ 8), event specific distress (IES-R), fatigue (FSI), sleep (ISI), well-being (MHC-SF), resilience (CD-RISC10), QOL (SF-20).

Tasso device blood collection for evaluation of inflammatory gene expression. Perform an active stand test Perform 6-minute walk

Post Intervention Visit (in person): collect within 1-2 weeks post intervention completion COMPASS-31: the composite autonomic symptom score Questionnaires: perceived stress (PSS), anxiety (GAD-7), depression (PHQ 8), event specific distress (IES-R), fatigue (FSI), sleep (ISI), well-being (MHC-SF), resilience (CD-RISC10), QOL (SF-20).

Tasso device blood collection for evaluation of inflammatory gene expression Perform an active stand test Perform Six-minute walk Three question mindfulness experience focused interview Frequency of Practice Logbook review

4-Week Post Intervention Visit (remote link / in person NOT required): collect 4 weeks (+2) post intervention Questionnaires: perceived stress (PSS), anxiety (GAD-7), depression (PHQ 8), event specific distress (IES-R), fatigue (FSI), sleep (ISI), well-being (MHC-SF), resilience (CD-RISC10), QOL (SF-20). 3-question Likert mindfulness experience survey

ELIGIBILITY:
Inclusion Criteria:

Adult females (18 years - 54 years of age)

* Previous SARS-CoV-2 infection confirmed by Polymerase chain reaction (PCR) testing and diagnoses of PASC and dysautonomia confirmed by objective testing (e.g., autonomic reflex screen, active stand test)
* Ability to comprehend English and complete assessments and patient-reported surveys
* Availability of a smartphone, tablet, or computer with Internet access

Exclusion Criteria:

* Inability to participate in the virtual intervention or complete outcomes surveys

  * Current participation regular mindfulness practice
  * Current enrollment in another COVID-19 related study.

Ages: 18 Years to 54 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2023-02-28 (Actual); Primary Completion 2023-07-29 (Actual); Study Completion 2023-07-29 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the composite autonomic symptom score COMPASS-31 for autonomic symptoms | Baseline / Pre Intervention(1-2 weeks prior to intervention), Post Intervention ( 1-2 weeks post intervention completion)
  COMPASS-31 (the composite autonomic symptom) score is a self-rating questionnaire evaluating six domains of autonomic function: orthostatic intolerance, vasomotor, secretomotor, gastrointestinal, bladder, and pupillomotor domains. The six domain scores sum to a total score of 0 to 100, and a higher score indicates more severe autonomic symptoms. It is based on the original Autonomic Symptom Profile (ASP) and COMPASS, is internally consistent and applies a much-simplified scoring algorithm suitable for widespread use in autonomic research and practice.
Change from baseline in Active Stand Test of hemodynamic symptom parameters, exercise tolerance. | Baseline / Pre Intervention(1-2 weeks prior to intervention), Post Intervention ( 1-2 weeks post intervention completion)
  Active Stand Test. Clinically, an active stand test can be used to assess short-term neural and cardiovascular function and identify the hemodynamic correlates of patient symptoms and attributable causes of (pre-)syncope, and to detect autonomic dysfunction, variants of orthostatic hypotension, postural orthostatic tachycardia syndrome and orthostatic hypertension. During a standardized active stand test procedure, heart rate and blood pressure are measured after resting lying down, then immediately upon standing and after 2, 5 and 10 minutes.
Change from baseline of Six Minute Walk in hemodynamic parameters, exercise tolerance | Baseline / Pre Intervention(1-2 weeks prior to intervention), Post Intervention ( 1-2 weeks post intervention completion)
  Six Minute Walk. The six-minute walk (6MWT) was developed in 1963 by Balke to evaluate functional capacity and endurance during physical activity. The standardized six-minute walk test (6MWT) measures the maximum distance an individual is able to walk over a total of six minutes. The individual is allowed to self-pace and rest as needed as they traverse back and forth along a flat marked walkway. Baseline heart rate and oxygen saturation are measured then continuously monitored to identify the lowest oxygen saturation, which may occur before the end of the test. The patient's baseline and post-test perceived dyspnea and fatigue are rated using the Borg scale 0-10 (0 none- 10 maximum).
Change from baseline in mean score in Health-Related Quality of Life (QOL) SF-20 | Baseline / Pre Intervention(1-2 weeks prior to intervention), Post Intervention (1-2 weeks post intervention completion); 4 weeks post intervention
  Self-reported QOL SF-20. A 20-item questionnaire. The survey measures health across 6 domains: physical functioning (6 questions), role functioning (2 questions), social functioning (1 question), mental health (5 questions), health perceptions (5 questions), and pain (1 question).
  Scores across each of these domains are reported on a 0% to 100% scale, with 0% representing the worst possible score in that domain and 100% the best possible score. Raw scores are transformed to fit the 0% to 100% interval as described in the original publication (note that for question #1 on general health, an initial transformation is performed as follows: 1 = 5, 2 = 4.36, 3 = 3.43, 4 = 1.99, 5 = 1). Reversal of scoring is completed as necessary such that the highest score always represents the best possible score. The exception to this scoring pattern is the pain score, for which 0% represents the best possible score and 100% the worst possible score.

SECONDARY OUTCOMES:
Change from baseline in mean scores of PSS- Perceived Stress Scale. | Baseline / Pre Intervention(1-2 weeks prior to intervention), Post Intervention (1-2 weeks post intervention completion); 4 weeks post intervention
  Perceived Stress Scale (PSS) appraises thoughts and feelings in perception of stress. It is a 10-item scale (score 0-40) with upper scores signifying increased perceived stress. While the aim is to capture stress level, the PSS is used to obtain a patients' perceptions of their own stress.
Change from baseline in mean scores of GAD7- Generalized Anxiety Disorder | Baseline / Pre Intervention(1-2 weeks prior to intervention), Post Intervention (1-2 weeks post intervention completion); 4 weeks post intervention
  Generalized Anxiety Disorder (GAD7) It is a 7-item scale (score 0-21), with acuity distinguished as mild (5-9), moderate (10-14) or severe (15-21) distress (Spitzer et al. 2006). The higher score indicates greater anxiety.
Change from baseline in mean scores of PHQ-8 - Depressive Symptoms | Baseline / Pre Intervention(1-2 weeks prior to intervention), Post Intervention (1-2 weeks post intervention completion); 4 weeks post intervention
  Depression (PHQ8) adapted from the PHQ-9, is established as a valid diagnostic and severity measure for depressive disorders in large clinical studies. A PHQ-8 score of 0 to 4 indicates no depression, of 5 to 9 indicates mild depression, of 10 to 14 indicates moderate depression, of 15 to 19 indicates moderately severe depression, and of 20 or higher indicates severe depression.
Change from baseline in mean scores of IES-R - event-related distress scale | Baseline / Pre Intervention(1-2 weeks prior to intervention), Post Intervention (1-2 weeks post intervention completion); 4 weeks post intervention
  Impact of Event Scale -Revised (IES-R). is a 22-item self-report measure that assesses subjective distress caused by traumatic events. The IES-R contains seven additional items related to the hyperarousal symptoms of PTSD, which were not included in the original IES. Items correspond directly to 14 of the 17 The Diagnostic and Statistical Manual of Mental Disorders (DSM-IV) symptoms of PTSD. Respondents are asked to identify a specific stressful life event and then indicate how much they were distressed or bothered during the past seven days by each "difficulty" listed. Items are rated on a 5-point scale ranging from 0 ("not at all") to 4 ("extremely"). The IES-R yields a total score (ranging from 0 to 88) and subscale scores can also be calculated for the Intrusion, Avoidance, and Hyperarousal subscales.
Change from baseline in mean scores of FSI - The Fatigue Symptom Inventory. | Baseline / Pre Intervention(1-2 weeks prior to intervention), Post Intervention (1-2 weeks post intervention completion); 4 weeks post intervention
  The Fatigue Symptom Inventory (FSI) is a 14-item self-report measure designed to assess the severity, frequency, and daily pattern of fatigue as well as its perceived interference with quality of life in the past week. Severity is measured on point scales (0=not at all fatigued; 10=as fatigued as I could be) that assess most, least, and average fatigue in the past week as well as current fatigue. Frequency is measured by the number of days (0-7) that respondents felt fatigued and the extent of each day they felt fatigued (0=none of the day; 10=the entire day). Perceived interference is measured on point scales (0=no interference; 10=extreme interference) that assess the degree to which fatigue was felt to interfere with with general level of activity, enjoyment, and mood.
Change from baseline in mean scores of the ISI - The Insomnia Severity Index | Baseline / Pre Intervention(1-2 weeks prior to intervention), Post Intervention (1-2 weeks post intervention completion); 4 weeks post intervention
  The Insomnia Severity Index (ISI) is a seven-item self-report questionnaire, which asks respondents to rate the nature and symptoms of their sleep problems. Dimensions evaluated are severity of sleep onset, sleep maintenance, and early morning awakening problems, sleep dissatisfaction, interference of sleep difficulties with daytime functioning, noticeability of sleep problems by others, and distress caused by the sleep difficulties. A 5-point Likert scale is used to rate each item (e.g., 0 = no problem; 4 = very severe problem), yielding a total score ranging from 0 to 28. The total score is interpreted as follows: absence of insomnia (0-7); sub-threshold insomnia (8-14); moderate insomnia (15-21); and severe insomnia (22-28).
Change from baseline in mean scores of well-being from MHC-SF-The Mental Health Continuum Short Form | Baseline / Pre Intervention(1-2 weeks prior to intervention), Post Intervention (1-2 weeks post intervention completion); 4 weeks post intervention
  The Mental Health Continuum Short Form (MHC-SF) is a 14- item scale containing 3 items for emotional (hedonic) well-being, 5 items for social well-being, and 6 items for psychological well-being (eudaimonic). Each of the items can be scored between 0 and 5, with the total score on the scale can range from 0 to 70 points. Higher scores indicate a higher level of emotional wellbeing. This scale also provides a flourishing and languishing mental health indicator based on these three subscales.
Change from baseline in mean scores of CD-RISC 10 - Connor Davidson Resilience Scale. | Baseline / Pre Intervention(1-2 weeks prior to intervention), Post Intervention (1-2 weeks post intervention completion); 4 weeks post intervention
  Connor Davidson Resilience Scale (CD-RISC 10) is a 10-item scale (score 0-40) that measures components of adaptation, coping and recovery in response to stressful events, trauma, or tragedy. The higher scores reflect greater resilience.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey J. Hsu, MD, PhD, Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA Health, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barizien N, Le Guen M, Russel S, Touche P, Huang F, Vallee A. Clinical characterization of dysautonomia in long COVID-19 patients. Sci Rep. 2021 Jul 7;11(1):14042. doi: 10.1038/s41598-021-93546-5. PMID 34234251
- [Background] Bisaccia G, Ricci F, Recce V, Serio A, Iannetti G, Chahal AA, Stahlberg M, Khanji MY, Fedorowski A, Gallina S. Post-Acute Sequelae of COVID-19 and Cardiovascular Autonomic Dysfunction: What Do We Know? J Cardiovasc Dev Dis. 2021 Nov 15;8(11):156. doi: 10.3390/jcdd8110156. PMID 34821709
- [Background] Raj SR, Arnold AC, Barboi A, Claydon VE, Limberg JK, Lucci VM, Numan M, Peltier A, Snapper H, Vernino S; American Autonomic Society. Long-COVID postural tachycardia syndrome: an American Autonomic Society statement. Clin Auton Res. 2021 Jun;31(3):365-368. doi: 10.1007/s10286-021-00798-2. Epub 2021 Mar 19. PMID 33740207
- [Background] Nalbandian A, Sehgal K, Gupta A, Madhavan MV, McGroder C, Stevens JS, Cook JR, Nordvig AS, Shalev D, Sehrawat TS, Ahluwalia N, Bikdeli B, Dietz D, Der-Nigoghossian C, Liyanage-Don N, Rosner GF, Bernstein EJ, Mohan S, Beckley AA, Seres DS, Choueiri TK, Uriel N, Ausiello JC, Accili D, Freedberg DE, Baldwin M, Schwartz A, Brodie D, Garcia CK, Elkind MSV, Connors JM, Bilezikian JP, Landry DW, Wan EY. Post-acute COVID-19 syndrome. Nat Med. 2021 Apr;27(4):601-615. doi: 10.1038/s41591-021-01283-z. Epub 2021 Mar 22. PMID 33753937
- [Background] Sykes DL, Holdsworth L, Jawad N, Gunasekera P, Morice AH, Crooks MG. Post-COVID-19 Symptom Burden: What is Long-COVID and How Should We Manage It? Lung. 2021 Apr;199(2):113-119. doi: 10.1007/s00408-021-00423-z. Epub 2021 Feb 11. PMID 33569660
- [Background] Sudre CH, Murray B, Varsavsky T, Graham MS, Penfold RS, Bowyer RC, Pujol JC, Klaser K, Antonelli M, Canas LS, Molteni E, Modat M, Jorge Cardoso M, May A, Ganesh S, Davies R, Nguyen LH, Drew DA, Astley CM, Joshi AD, Merino J, Tsereteli N, Fall T, Gomez MF, Duncan EL, Menni C, Williams FMK, Franks PW, Chan AT, Wolf J, Ourselin S, Spector T, Steves CJ. Attributes and predictors of long COVID. Nat Med. 2021 Apr;27(4):626-631. doi: 10.1038/s41591-021-01292-y. Epub 2021 Mar 10. PMID 33692530
- [Background] Antonova E, Schlosser K, Pandey R, Kumari V. Coping With COVID-19: Mindfulness-Based Approaches for Mitigating Mental Health Crisis. Front Psychiatry. 2021 Mar 23;12:563417. doi: 10.3389/fpsyt.2021.563417. eCollection 2021. PMID 33833695
- [Background] Blanck P, Perleth S, Heidenreich T, Kroger P, Ditzen B, Bents H, Mander J. Effects of mindfulness exercises as stand-alone intervention on symptoms of anxiety and depression: Systematic review and meta-analysis. Behav Res Ther. 2018 Mar;102:25-35. doi: 10.1016/j.brat.2017.12.002. Epub 2017 Dec 20. PMID 29291584
- [Background] Deng J, Zhou F, Hou W, Silver Z, Wong CY, Chang O, Huang E, Zuo QK. The prevalence of depression, anxiety, and sleep disturbances in COVID-19 patients: a meta-analysis. Ann N Y Acad Sci. 2021 Feb;1486(1):90-111. doi: 10.1111/nyas.14506. Epub 2020 Oct 2. PMID 33009668
- [Background] Johansson M, Stahlberg M, Runold M, Nygren-Bonnier M, Nilsson J, Olshansky B, Bruchfeld J, Fedorowski A. Long-Haul Post-COVID-19 Symptoms Presenting as a Variant of Postural Orthostatic Tachycardia Syndrome: The Swedish Experience. JACC Case Rep. 2021 Apr;3(4):573-580. doi: 10.1016/j.jaccas.2021.01.009. Epub 2021 Mar 10. PMID 33723532
- [Background] Graham EL, Clark JR, Orban ZS, Lim PH, Szymanski AL, Taylor C, DiBiase RM, Jia DT, Balabanov R, Ho SU, Batra A, Liotta EM, Koralnik IJ. Persistent neurologic symptoms and cognitive dysfunction in non-hospitalized Covid-19 "long haulers". Ann Clin Transl Neurol. 2021 May;8(5):1073-1085. doi: 10.1002/acn3.51350. Epub 2021 Mar 30. PMID 33755344
- [Background] Johns SA, Tarver WL, Secinti E, Mosher CE, Stutz PV, Carnahan JL, Talib TL, Shanahan ML, Faidley MT, Kidwell KM, Rand KL. Effects of mindfulness-based interventions on fatigue in cancer survivors: A systematic review and meta-analysis of randomized controlled trials. Crit Rev Oncol Hematol. 2021 Apr;160:103290. doi: 10.1016/j.critrevonc.2021.103290. Epub 2021 Mar 4. PMID 33675902
- [Background] Mazza MG, De Lorenzo R, Conte C, Poletti S, Vai B, Bollettini I, Melloni EMT, Furlan R, Ciceri F, Rovere-Querini P; COVID-19 BioB Outpatient Clinic Study group; Benedetti F. Anxiety and depression in COVID-19 survivors: Role of inflammatory and clinical predictors. Brain Behav Immun. 2020 Oct;89:594-600. doi: 10.1016/j.bbi.2020.07.037. Epub 2020 Jul 30. PMID 32738287
- [Background] Pascoe MC, Thompson DR, Jenkins ZM, Ski CF. Mindfulness mediates the physiological markers of stress: Systematic review and meta-analysis. J Psychiatr Res. 2017 Dec;95:156-178. doi: 10.1016/j.jpsychires.2017.08.004. Epub 2017 Aug 23. PMID 28863392
- [Background] Pascoe MC, de Manincor M, Tseberja J, Hallgren M, Baldwin PA, Parker AG. Psychobiological mechanisms underlying the mood benefits of meditation: A narrative review. Compr Psychoneuroendocrinol. 2021 Mar 10;6:100037. doi: 10.1016/j.cpnec.2021.100037. eCollection 2021 May. PMID 35757358
- [Background] Spijkerman MP, Pots WT, Bohlmeijer ET. Effectiveness of online mindfulness-based interventions in improving mental health: A review and meta-analysis of randomised controlled trials. Clin Psychol Rev. 2016 Apr;45:102-14. doi: 10.1016/j.cpr.2016.03.009. Epub 2016 Apr 1. PMID 27111302
- [Background] Simonelli C, Paneroni M, Vitacca M, Ambrosino N. Measures of physical performance in COVID-19 patients: a mapping review. Pulmonology. 2021 Nov-Dec;27(6):518-528. doi: 10.1016/j.pulmoe.2021.06.005. Epub 2021 Jun 24. PMID 34284976
- [Background] Zhang D, Lee EKP, Mak ECW, Ho CY, Wong SYS. Mindfulness-based interventions: an overall review. Br Med Bull. 2021 Jun 10;138(1):41-57. doi: 10.1093/bmb/ldab005. PMID 33884400
- [Background] Zou L, Sasaki JE, Zeng N, Wang C, Sun L. A Systematic Review With Meta-Analysis of Mindful Exercises on Rehabilitative Outcomes Among Poststroke Patients. Arch Phys Med Rehabil. 2018 Nov;99(11):2355-2364. doi: 10.1016/j.apmr.2018.04.010. Epub 2018 May 5. PMID 29738744
- [Background] Bower JE, Crosswell AD, Stanton AL, Crespi CM, Winston D, Arevalo J, Ma J, Cole SW, Ganz PA. Mindfulness meditation for younger breast cancer survivors: a randomized controlled trial. Cancer. 2015 Apr 15;121(8):1231-40. doi: 10.1002/cncr.29194. Epub 2014 Dec 23. PMID 25537522
- [Background] Boyle CC, Cole SW, Dutcher JM, Eisenberger NI, Bower JE. Changes in eudaimonic well-being and the conserved transcriptional response to adversity in younger breast cancer survivors. Psychoneuroendocrinology. 2019 May;103:173-179. doi: 10.1016/j.psyneuen.2019.01.024. Epub 2019 Jan 23. PMID 30703712
- [Background] Tawakol A, Ishai A, Takx RA, Figueroa AL, Ali A, Kaiser Y, Truong QA, Solomon CJ, Calcagno C, Mani V, Tang CY, Mulder WJ, Murrough JW, Hoffmann U, Nahrendorf M, Shin LM, Fayad ZA, Pitman RK. Relation between resting amygdalar activity and cardiovascular events: a longitudinal and cohort study. Lancet. 2017 Feb 25;389(10071):834-845. doi: 10.1016/S0140-6736(16)31714-7. Epub 2017 Jan 12. PMID 28088338
- [Background] Scott-Sheldon LAJ, Gathright EC, Donahue ML, Balletto B, Feulner MM, DeCosta J, Cruess DG, Wing RR, Carey MP, Salmoirago-Blotcher E. Mindfulness-Based Interventions for Adults with Cardiovascular Disease: A Systematic Review and Meta-Analysis. Ann Behav Med. 2020 Jan 1;54(1):67-73. doi: 10.1093/abm/kaz020. PMID 31167026
- [Background] Shaygan M, Yazdani Z, Valibeygi A. The effect of online multimedia psychoeducational interventions on the resilience and perceived stress of hospitalized patients with COVID-19: a pilot cluster randomized parallel-controlled trial. BMC Psychiatry. 2021 Feb 11;21(1):93. doi: 10.1186/s12888-021-03085-6. PMID 33573631
- [Background] O'Donnell KT, Dunbar M, Speelman DL. Effectiveness of using a meditation app in reducing anxiety and improving well-being during the COVID-19 pandemic: A structured summary of a study protocol for a randomized controlled trial. Trials. 2020 Dec 9;21(1):1006. doi: 10.1186/s13063-020-04935-6. PMID 33298117
- [Background] Kubo A, Kurtovich E, McGinnis M, Aghaee S, Altschuler A, Quesenberry C Jr, Kolevska T, Liu R, Greyz-Yusupov N, Avins A. Pilot pragmatic randomized trial of mHealth mindfulness-based intervention for advanced cancer patients and their informal caregivers. Psychooncology. 2024 Feb;33(2):e5557. doi: 10.1002/pon.5557. Epub 2020 Oct 5. PMID 32979294
- [Background] Levine GN, Lange RA, Bairey-Merz CN, Davidson RJ, Jamerson K, Mehta PK, Michos ED, Norris K, Ray IB, Saban KL, Shah T, Stein R, Smith SC Jr; American Heart Association Council on Clinical Cardiology; Council on Cardiovascular and Stroke Nursing; and Council on Hypertension. Meditation and Cardiovascular Risk Reduction: A Scientific Statement From the American Heart Association. J Am Heart Assoc. 2017 Sep 28;6(10):e002218. doi: 10.1161/JAHA.117.002218. PMID 28963100
- [Background] Campbell-Sills L, Stein MB. Psychometric analysis and refinement of the Connor-davidson Resilience Scale (CD-RISC): Validation of a 10-item measure of resilience. J Trauma Stress. 2007 Dec;20(6):1019-28. doi: 10.1002/jts.20271. PMID 18157881
- [Background] Cohen S, Kamarck T, Mermelstein R. A global measure of perceived stress. J Health Soc Behav. 1983 Dec;24(4):385-96. No abstract available. PMID 6668417
- [Background] Finucane C, van Wijnen VK, Fan CW, Soraghan C, Byrne L, Westerhof BE, Freeman R, Fedorowski A, Harms MPM, Wieling W, Kenny R. A practical guide to active stand testing and analysis using continuous beat-to-beat non-invasive blood pressure monitoring. Clin Auton Res. 2019 Aug;29(4):427-441. doi: 10.1007/s10286-019-00606-y. Epub 2019 May 10. PMID 31076939
- [Background] Keyes CL, Wissing M, Potgieter JP, Temane M, Kruger A, van Rooy S. Evaluation of the mental health continuum-short form (MHC-SF) in setswana-speaking South Africans. Clin Psychol Psychother. 2008 May-Jun;15(3):181-92. doi: 10.1002/cpp.572. PMID 19115439
- [Background] Kroenke K, Strine TW, Spitzer RL, Williams JB, Berry JT, Mokdad AH. The PHQ-8 as a measure of current depression in the general population. J Affect Disord. 2009 Apr;114(1-3):163-73. doi: 10.1016/j.jad.2008.06.026. Epub 2008 Aug 27. PMID 18752852
- [Background] Sletten DM, Suarez GA, Low PA, Mandrekar J, Singer W. COMPASS 31: a refined and abbreviated Composite Autonomic Symptom Score. Mayo Clin Proc. 2012 Dec;87(12):1196-201. doi: 10.1016/j.mayocp.2012.10.013. PMID 23218087
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Weiss, D. S., & Marmar, C. R. (1996). The Impact of Event Scale - Revised. In J. Wilson & T. M. Keane (Eds.), Assessing psychological trauma and PTSD (pp. 399-411). New York: Guilford.
- [Background] BALKE B. A SIMPLE FIELD TEST FOR THE ASSESSMENT OF PHYSICAL FITNESS. REP 63-6. Rep Civ Aeromed Res Inst US. 1963 Apr:1-8. No abstract available. PMID 14131272
- [Background] Hann DM, Jacobsen PB, Azzarello LM, Martin SC, Curran SL, Fields KK, Greenberg H, Lyman G. Measurement of fatigue in cancer patients: development and validation of the Fatigue Symptom Inventory. Qual Life Res. 1998 May;7(4):301-10. doi: 10.1023/a:1024929829627. PMID 9610214
- [Background] Bastien CH, Vallieres A, Morin CM. Validation of the Insomnia Severity Index as an outcome measure for insomnia research. Sleep Med. 2001 Jul;2(4):297-307. doi: 10.1016/s1389-9457(00)00065-4. PMID 11438246
- [Background] Stewart AL, Hays RD, Ware JE Jr. The MOS short-form general health survey. Reliability and validity in a patient population. Med Care. 1988 Jul;26(7):724-35. doi: 10.1097/00005650-198807000-00007. No abstract available. PMID 3393032